CLINICAL TRIAL: NCT05957068
Title: Breast Cancer Exercise Intervention Study (BREXINT)
Brief Title: Breast Cancer Exercise Intervention Study
Acronym: BREXINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Singapore Cancer Society (Other); Genome Institute of Singapore (Other); National University of Singapore (Other); Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BREXINT
Record Dates: First submitted 2023-06-13; First posted 2023-07-24 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Early-stage Breast Cancer; Locally Advanced Breast Cancer
Keywords: BREXINT; Muscular Strength; Cardiorespiratory Fitness; Quality of Life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomised into 2 groups: exercise (intervention group, N = 1078) and usual care (control group, N = 1078). The exercise intervention group will undergo an aerobic exercise and strength training programme.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): The exercise intervention group will undergo an aerobic exercise and strength training programme, comprising 3 sessions per week, spanning 24 weeks (total: 3x24=72 sessions).
  Interventions: Behavioral: Exercise Programme
- Control (Experimental): The usual care group.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Exercise Programme — Aerobic exercise consists of 20-minute brisk walks or jogs (5-6 km/h) on the treadmill each session, reaching a heart rate corresponding to 50%-70% of the patient's VO2max (VO2max is determined before embarking on the exercise programme). Study participants are expected to aim for 50% VO2max at the start of the exercise programme, and gradually increasing to 70% VO2max in subsequent exercise sessions. Strength training comprises a series of circuit resistance exercises targeting the major muscle groups. Patients will perform 2-4 sets of these exercises each session, 8-10 repetitions per set. Both aerobic exercise and strength training are done in the same session. With warm-up and cool-down, each session is estimated to take up 1 hour.
  Arms: Exercise
Behavioral: Control — Usual care group.
  Arms: Control

SUMMARY:
This is a 24-week exercise programme consisting of aerobic exercise and muscle strength training, 3 sessions per week. The first 9 sessions are supervised by physiotherapists in person, followed by 63 sessions monitored remotely (video) or supervised by trainers at ActiveSG (Sport Singapore) gyms.

DETAILED DESCRIPTION:
This is a multi-centre, randomised controlled study of a 6-month (24-week) exercise programme versus observation in 2156 early stage and locally advanced breast cancer patients who have undergone curative breast surgery, and who have completed (neo)adjuvant chemotherapy (if given) or radiotherapy (if given). Patients are stratified by centre (NCC/SGH, NUH), menopausal status, ER/PR status, body fat/muscle ratio.

Cardiorespiratory fitness, muscle strength, level of routine daily physical activity, body fat/muscle ratio are monitored during the study period.

Blood is collected at baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks, then annually for 4 times.

Questionnaires are periodically conducted to assess quality of life (QoL). A food diary is kept.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically proven stage 1, 2, or 3 breast cancer
* Patients who have undergone curative breast surgery
* Patients who have received (neo)adjuvant chemotherapy (if given) and/or radiotherapy (if given)
* Females aged 21 years and older
* ≤ 8 weeks from breast surgery, or the last adjuvant chemotherapy or radiotherapy session, whichever is latest.

Exclusion Criteria:

* Cardiovascular, respiratory, musculoskeletal problems that preclude moderate physical activity.
* Major medical problems that are deemed by the investigator to be unsuitable for enrollment.

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2156 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2033-05-31 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | Up to 5 years.
  From the date of randomization to when an event, i.e. relapse, has occurred.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 5 years.
  From the date of randomization to when an event, i.e. death, has occurred.

OTHER OUTCOMES:
Body fat/muscle ratio. | Week 0, Week 8, Week 16 and Week 24.
  Body fat mass (in grams) divided by body muscle mass (in grams).
Changes in absolute and relative VO2. | Week 8, Week 16 and Week 24.
  Changes in absolute (L/min) and relative VO2 (mL/kg/min) at 8, 16 and 24 weeks from baseline.
Changes in heart rate at rest and during CPET. | Week 8, Week 16 and Week 24.
  Changes in heart rate (HR, beats/min) at rest and during CPET, at 8, 16 and 24 weeks from baseline.
Changes in oxygen pulse (VO2/HR) during CPET. | Week 8, Week 16 and Week 24.
  Changes in oxygen pulse (VO2/HR) during CPET, at 8, 16, and 24 weeks from baseline.
Changes in respiratory exchange ratio (RER) during CPET. | Week 8, Week 16 and Week 24.
  Changes in respiratory exchange ratio (RER, unitless) during CPET, at 8, 16, and 24 weeks from baseline
Changes in weight lifted 10 repetition maximum. | Week 0, Week 8, Week 16 and Week 24.
  Changes in weight lifted 10 repetition maximum (10-RM, Kg) for: a. Chest press; b. Latissimus pull-down; c. 2-arm curl; and d. Leg press.
Changes in absolute fat mass and relative fat mass from baseline. | Week 8, Week 16 and Week 24.
  Changes in absolute fat mass (kg) and relative fat mass (%) at 8, 16, and 24 weeks from baseline.
Changes in absolute lean mass and relative lean mass from baseline. | Week 8, Week 16 and Week 24.
  Changes in absolute lean mass (kg) and relative lean mass (%) at 8, 16, and 24 weeks from baseline.
Changes in absolute and relative bone mineral density (BMD) at 8, 16, and 24 weeks from baseline. | Week 8, Week 16 and Week 24.
  Changes in absolute and relative bone mineral density (BMD, in g/cm^2) at 8, 16, and 24 weeks from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Elaine LIM, MD, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (3):
- Singapore (3):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Once data is available, only de-identified IPD will be shared to collaborators.